CLINICAL TRIAL: NCT00549939
Title: 12-week, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Investigate the Efficacy, Pharmacodynamic and Safety of 2 Doses of Alfuzosin (0.1 mg/kg/Day, 0.2 mg/kg/Day) in the Treatment of Children and Adolescents 2-16 Years With Elevated Detrusor Leak Point Pressure of Neuropathic Etiology Followed by a 40-week Open-label Extension
Brief Title: Alfuzosin Treatment in Children and Adolescents With Neurogenic Urinary Bladder Dysfunction
Acronym: ALFACHIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC5722; 2004-002397-38 (EudraCT Number)
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Results first posted 2011-02-08 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Neurogenic Urinary Bladder
Keywords: child; bladder; neuropathic; alpha blockers
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo 0.1 mg/kg/day or 0.2 mg/kg/day
  Interventions: Drug: Placebo
- Alfuzosin 0.1 mg/kg/day (Experimental)
  Interventions: Drug: Alfuzosin
- Alfuzosin 0.2 mg/kg/day (Experimental)
  Interventions: Drug: Alfuzosin

INTERVENTIONS:
Drug: Alfuzosin — Form: solution or tablet according to age
  Route: oral
  Dose: daily dose adjusted to body weight
  Other Names: SL770499
  Arms: Alfuzosin 0.1 mg/kg/day; Alfuzosin 0.2 mg/kg/day
Drug: Placebo — Form: matching solution or matching tablet according to age
  Route: oral
  Dose: daily dose adjusted to body weight
  Arms: Placebo

SUMMARY:
The primary objective of the study was to evaluate the efficacy of Alfuzosin in comparison to Placebo on the detrusor Leak Point Pressure (LPP) in children and adolescents 2-16 years of age with elevated detrusor LPP of neuropathic etiology and detrusor LPP ≥ 40 cm H2O.

Secondary objectives were:

* To investigate the safety and tolerability of two doses of Alfuzosin in comparison to Placebo in children and adolescents,
* To evaluate the effects of the two doses of Alfuzosin in comparison to Placebo on:

  * Detrusor compliance,
  * Urinary tract infection,
* To investigate the pharmacokinetics of Alfuzosin (population kinetics),
* To evaluate the 12-month long-term safety of Alfuzosin 0.1 mg/kg/day and 0.2 mg/kg/day.

The study consisted of 2 periods:

* a 12-week double blind treatment period where patients were to receive either Alfuzosin 0.1 mg/kg/day or Alfuzosin 0.2 mg/kg/day or placebo then,
* a 40-week open label extension treatment period where patients were to receive either Alfuzosin 0.1 mg/kg/day or Alfuzosin 0.2 mg/kg/day.

DETAILED DESCRIPTION:
Patients who met the study entry criteria were randomized (2:1:2:1) to one of the 4 dosage groups (Alfuzosin 0.1 mg/kg/day, matching placebo 0.1 mg/kg/day, Alfuzosin 0.2 mg/mg/kg, matching placebo 0.2 mg/kg/day).

Patients received their treatment using either solution or tablet formulation depending on age as follows:

* Solution to children 2-7 years of age or, children and adolescents 8-16 years of age if they were unable to swallow tablets or they preferred to take the solution or if they had a body weight < 30kg. The daily dose was devided in 3 doses given at at breakfast, lunch and dinner.
* Tablet to children and adolescents 8-16 years of age who were able to swallow tablets and had a body weight ≥ 30kg. The daily dose was devided in 2 doses given at at breakfast and dinner.

Patients who have completed the 12-week double-blind phase were offered to continue in the 40-week open-label extension study.

* Patients receiving Alfuzosin continued with their dosing regimen.
* Patients receiving Placebo were switched to Alfuzosin with a dose corresponding to their randomization dose group.

All patients had a one-week follow-up period after last dose intake.

ELIGIBILITY:
Inclusion Criteria:

* Patient with elevated detrusor Leak Point Pressure (LPP) of neuropathic etiology and Detrusor LPP ≥ 40 cm H2O and < 100 cm H2O.

Exclusion Criteria:

* Urological surgery in the last 4 months prior to the study,
* Patients who have urethral dilatation in the last 3 months prior to the baseline urodynamic assessment,
* α-blocker therapy in the last 4 weeks prior to the baseline urodynamic assessment,
* Detrusor injections of botulinum toxin in the last 6 months,
* Urological diseases/conditions other than functional bladder obstruction of neuropathic etiology that can lead to upper urinary tract dilatation (e.g., bladder anomalies, ureterocele),
* History of intolerance to α-blocker therapy,
* Orthostatic hypotension,
* History of risk factors for Torsade de pointes (e.g., family history of Long QT Syndrome).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (18):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Aministrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Belgrade, Serbia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 55 sites in 18 countries. A total of 261 patients were screened between September 2007 and November 2008.
Pre-assignment Details: 172/261 patients were randomized in the 12-week double blind phase.
  89/261 patients were not randomized for the following reasons:
  * Adverse event (1 patient*),
  * Inclusion/Exclusion criteria not met (69 patients*),
  * Subject's request (11 patients*),
  * Other (13 patients*).
  '*' Patients could have several reasons.
Groups:
- Placebo: Alfuzosin 0.1 mg/kg/day matching placebo or Alfuzosin 0.2 mg/kg/day matching placebo
Period: 12-week Double Blind Treatment Period
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Started | 57 (29 (Alfuzosin 0.1 mg/kg/day matching placebo) + 28 (Alfuzosin 0.2 mg/kg/day matching placebo)) | 57 | 58
Completed | 56 | 55 | 56
Not Completed | 1 | 2 | 2
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Too many blood draws | 0 | 1 | 0
Period: 40-week Open Label Treatment Period
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Started | 0 (54 patients continued and switched to Alfuzosin: 26 to 0.1 mg/kg/day and 28 to 0.2 mg/kg/day.) | 80 (54 patients continued Alfuzosin 0.1 mg/kg/day and 26 patients started Alfuzosin 0.1 mg/kg/day.) | 83 (55 patients continued Alfuzosin 0.2 mg/kg/day and 28 patients started Alfuzosin 0.2 mg/kg/day.)
Completed | 0 | 75 | 78
Not Completed | 0 | 5 | 5
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Other | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day | Total
Number analyzed (Participants) | 57 | 57 | 58 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (4.4) | 7.9 (3.9) | 8.7 (3.9) | 8.3 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 30 | 85
  Male | 29 | 30 | 28 | 87
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 5 | 18
  Portugal | 2 | 1 | 3 | 6
  Serbia | 4 | 6 | 7 | 17
  Taiwan | 0 | 1 | 1 | 2
  Estonia | 1 | 1 | 1 | 3
  Slovakia | 6 | 7 | 1 | 14
  Spain | 2 | 3 | 2 | 7
  Turkey | 1 | 2 | 3 | 6
  Russian Federation | 8 | 7 | 4 | 19
  India | 2 | 9 | 9 | 20
  France | 1 | 2 | 4 | 7
  Canada | 3 | 1 | 2 | 6
  Malaysia | 3 | 0 | 0 | 3
  Poland | 15 | 10 | 14 | 39
  Germany | 3 | 0 | 2 | 5
Urinary Tract Infection (UTI) history in the last 3 months [Number; unit: participants]
  No UTI episode | 48 | 50 | 40 | 138
  One UTI episode | 8 | 5 | 16 | 29
  Two UTI episodes | 1 | 2 | 2 | 5
Study drug formulation [Number; unit: participants]
  Solution (2-7 years) | 28 | 28 | 28 | 84
  Solution (8-16 years) | 8 | 10 | 9 | 27
  Tablets (8-16 years) | 21 | 19 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Detrusor Leak Point Pressure (LPP) < 40 cm H2O
Description: Detrusor Leak Point Pressure (LPP) was measured by cystometry.
  For each measure, 2 or 3 cystometries were carried out depending on the difference between the 2 first LPP values (if the difference ≥ 20 cm H2O, a 3rd cystometry was done). The lowest value was retained.
  Investigators reading was then consolidated by the review of all cystometry data by 2 external "Expert Reviewers", who were blinded for the study treatment.
  The analysis was performed on consolidated investigators data (i.e. endorsed by the Investigator taking into account reviewers opinion).
Time Frame: 12 weeks (double blind treatment period)
Population: The Intent-to-treat (ITT) population was used for the analysis. All randomized patients were included in the analysis in the treatment group to which they were allocated as per randomization.
Measure: Number; unit: participants
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 57 | 57 | 58
participants
  < 40 cmH2O ("Success") | 23 | 23 | 28
  ≥ 40 cmH2O or missing ("Failure") | 34 | 34 | 30
Statistical Analysis 1: Comparison: Placebo vs Alfuzosin 0.1 mg/kg/Day; Test type: Superiority or Other; p = 1.00, Fisher Exact — P-value was adjusted for multiplicity using the Hochberg procedure. The a priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Placebo vs Alfuzosin 0.2 mg/kg/Day; Test type: Superiority or Other; p = 0.91, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Detrusor Leak Point Pressure (LPP)
Description: Detrusor Leak Point Pressure (LPP) was assessed at baseline and 12 weeks as described for the primary outcome measure.
Time Frame: baseline and 12 weeks (double blind treatment period)
Population: The analysis was performed on the Intent-to-treat (ITT) population excluding the patients who didn't have baseline and/or post-baseline LPP values. Patients were included in the treatment group to which they were allocated as per randomization.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 54 | 53 | 56
cmH2O
  Baseline | 54.2 (12.6) | 53.3 (13.4) | 50.9 (10.0)
  12 Weeks | 48.2 (23.4) | 41.6 (18.2) | 39.4 (19.5)

3. Secondary Outcome: Absolute Change in Detrusor LPP
Description: Absolute change = Detrusor LPP at 12 weeks - Detrusor LPP at baseline
Time Frame: 12 weeks ((double blind treatment period)
Population: The analysis was performed on the same population as previously (i.e. ITT population excluding the patients who didn't have baseline and/or post-baseline value).
Measure: Least Squares Mean (Standard Error); unit: cmH2O
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 54 | 53 | 56
cmH2O | -5.4 (2.8) | -11.7 (2.8) | -12.5 (2.8)
Statistical Analysis 1: Comparison: Placebo vs Alfuzosin 0.1 mg/kg/Day; Change in detrusor LPP was analyzed using a three-way analysis of covariance (ANCOVA) including 3 variables as fixed effects: * treatment group (alfuzosin 0.1 mg/kg/day, alfuzosin 0.2 mg/kg/day or placebo), * age/formulation group (2-7 years of age on solution, 8-16 years of age on solution or 8-16 years of age on tablets), * anticholinergic/antimuscarinic use (yes or no), and using centered baseline detrusor LPP as covariate; Test type: Superiority or Other; p = 0.1040, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference versus Placebo = -6.2, 95% CI 2-sided [-13.72 to 1.29], Standard Error of Mean 3.80
Statistical Analysis 2: Comparison: Placebo vs Alfuzosin 0.2 mg/kg/Day; Test type: Superiority or Other; p = 0.1040, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference versus Placebo = -7.1, 95% CI 2-sided [-14.51 to 0.39], Standard Error of Mean 3.77

4. Secondary Outcome: Relative Change in Detrusor LPP
Description: Relative change = 100 * (Detrusor LPP at 12 weeks - Detrusor LPP at baseline) / Detrusor LPP at baseline
Time Frame: 12 weeks (double blind treatment period)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of cmH2O
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 54 | 53 | 56
percentage of cmH2O | -9.2 (5.53) | -20.6 (5.56) | -23.5 (5.51)
Statistical Analysis 1: Comparison: Placebo vs Alfuzosin 0.1 mg/kg/Day; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1338, ANCOVA — P-values was adjusted for multiplicity using the Hochberg procedure. The a priori threshold for statistical significance was 0.05; LS Mean difference versus Placebo = -11.4, 95% CI 2-sided [-26.27 to 3.53], Standard Error of Mean 7.54
Statistical Analysis 2: Comparison: Placebo vs Alfuzosin 0.2 mg/kg/Day; Test type: Superiority or Other; p = 0.1152, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference versus Placebo = -14.3, 95% CI 2-sided [-29.10 to 0.47], Standard Error of Mean 7.48

5. Secondary Outcome: Detrusor Compliance
Description: Detrusor compliance is defined as the relationship between change in detrusor volume and change in detrusor pressure.
  It was calculated by dividing the volume change (ΔV) by the change in detrusor pressure (Δpdet) during that change in detrusor volume at leak point (C= ΔV/Δpdet).
Time Frame: baseline and 12 weeks (double blind treatment period)
Population: The analysis was performed on the intent-to-treat (ITT) population excluding the patients who didn't have baseline and/or post baseline detrusor compliance values. Patients were included in the treatment group to which they were allocated as per randomization.
Measure: Mean (Standard Deviation); unit: mL/cmH20
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 54 | 52 | 55
mL/cmH20
  Baseline | 3.4 (2.8) | 3.4 (2.8) | 3.3 (2.5)
  12 weeks | 4.8 (5.0) | 5.3 (4.9) | 5.8 (5.9)

6. Secondary Outcome: Relative Change in Detrusor Compliance
Description: Relative change = 100 * (Detrusor compliance at 12 weeks - Detrusor compliance at baseline) / Detrusor compliance at baseline
Time Frame: 12 weeks (double blind treatment period)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of mL/cmH2O
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 54 | 52 | 55
percentage of mL/cmH2O | 113.6 (35.26) | 126.6 (35.76) | 98.6 (35.24)
Statistical Analysis 1: Comparison: Placebo vs Alfuzosin 0.1 mg/kg/Day; Change in detrusor compliance was analyzed using a three-way analysis of covariance (ANCOVA) including 3 variables as fixed effects: * treatment group (alfuzosin 0.1 mg/kg/day, alfuzosin 0.2 mg/kg/day or placebo), * age/formulation group (2-7 years of age on solution, 8-16 years of age on solution or 8-16 years of age on tablets), * anticholinergic/antimuscarinic use (yes or no), and using centered baseline detrusor compliance as covariate; Test type: Superiority or Other; p = 0.7889, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alfuzosin 0.2 mg/kg/Day; Test type: Superiority or Other; p = 0.7889, ANCOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Symptomatic Urinary Tract Infection (UTI) Episodes
Description: When a patient presented with symptoms such as pain, fever or hematuria (discretion of the Investigator), an urinalysis was performed including a dipstick and a quantitative urine culture.
  A symptomatic UTI was defined as the presence of symptoms and a positive culture with > 100 000 Colony Forming Units (CFUs) with a single organism.
Time Frame: 12 weeks (double blind treatment period)
Population: The analysis was performed on the intent-to-treat (ITT) population. All randomized patients were included in the analysis in the treatment group to which they were allocated as per randomization.
Measure: Number; unit: participants
Arm/Group | Placebo | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 57 | 57 | 58
participants
  No symptomatic UTI | 50 | 53 | 51
  One symptomatic UTI | 5 | 3 | 6
  Two symptomatic UTI | 2 | 1 | 1

8. Secondary Outcome: Number of Participants With Symptomatic Urinary Tract Infection (UTI) Episodes
Description: Symptomatic UTI episodes were assessed similar to the previous outcome measure but for a longer follow-up period.
Time Frame: 52 weeks (double blind treatment period + open label extension treatment period)
Population: The analysis was performed on the exposed population (i.e. all patients who received at least one dose of Alfuzosin regardless of the amount of treatment received). It included 3 + 3 patients treated during the 1st treatment period only, 26 + 28 patients treated during the 2nd treatment period only and 54 + 55 patients treated during both periods.
Measure: Number; unit: participants
Arm/Group | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Number analyzed (Participants) | 83 | 86
participants
  No symptomatic UTI | 66 | 70
  One symptomatic UTI | 12 | 13
  Two symptomatic UTI | 3 | 0
  Three symptomatic UTI | 1 | 1
  Four symptomatic UTI | 1 | 2

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) regardless of seriousness or relationship to drug, spanning from signature of the Informed Consent Form up to the last visit were collected.
Description: The analysis was performed on the exposed population (i.e. all patients who received at least one dose of Alfuzosin, whatever the study period and regardless of the amount of treatment received) and included all AE that developed/worsened during the 'on treatment period' (i.e. from first dose up to 2 days after the last dose).
Arm/Group | Alfuzosin 0.1 mg/kg/Day | Alfuzosin 0.2 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 10/83 | 7/86
Other Adverse Events (participants affected / at risk) | 37/83 | 43/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alfuzosin 0.1 mg/kg/Day (N=83) | Alfuzosin 0.2 mg/kg/Day (N=86)
VIRAL INFECTION (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 1
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 2 | 0
TETHERED CORD SYNDROME (Nervous system disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0
URETHRAL HAEMORRHAGE (Renal and urinary disorders) | 1 | 0
ARNOLD-CHIARI MALFORMATION (Congenital, familial and genetic disorders) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
VENTRICULOPERITONEAL SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alfuzosin 0.1 mg/kg/Day (N=83) | Alfuzosin 0.2 mg/kg/Day (N=86)
NASOPHARYNGITIS (Infections and infestations) | 6 | 12
CYSTITIS (Infections and infestations) | 5 | 9
URINARY TRACT INFECTION (Infections and infestations) | 9 | 6
PHARYNGITIS (Infections and infestations) | 8 | 5
RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 5
DIARRHOEA (Gastrointestinal disorders) | 8 | 10
VOMITING (Gastrointestinal disorders) | 4 | 6
PYREXIA (General disorders) | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the investigators can publish the results. Prior to publication, the sponsor shall review the manuscript and can request changes, provided they do not jeopardize the accuracy and/or the scientific value of the publication. The approval is given in writing by the sponsor, not to exceed 90 days.

To protect by a property right any information the sponsor can postpone the publication, for a period not to exceed 18 months.